CLINICAL TRIAL: NCT04269837
Title: Counseling Intervention During Radiation Therapy for Women With Gynecologic Cancer
Brief Title: Sexual Health Counseling Intervention During Radiation Therapy in Improving Quality of Life for Women With Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Allison Quick, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-19322; NCI-2020-00135 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Malignant Female Reproductive System Neoplasm; Stage I Cervical Cancer AJCC v8; Stage I Uterine Corpus Cancer AJCC v8; Stage I Vaginal Cancer AJCC v8; Stage I Vulvar Cancer AJCC v8; Stage IA Cervical Cancer AJCC v8; Stage IA Uterine Corpus Cancer AJCC v8; Stage IA Vaginal Cancer AJCC v8; Stage IA Vulvar Cancer AJCC v8; Stage IA1 Cervical Cancer AJCC v8; Stage IA2 Cervical Cancer AJCC v8; Stage IB Cervical Cancer AJCC v8; Stage IB Uterine Corpus Cancer AJCC v8; Stage IB Vaginal Cancer AJCC v8; Stage IB Vulvar Cancer AJCC v8; Stage IB1 Cervical Cancer AJCC v8; Stage IB2 Cervical Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage II Uterine Corpus Cancer AJCC v8; Stage II Vaginal Cancer AJCC v8; Stage II Vulvar Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA Vaginal Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage IIB Vaginal Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage III Vaginal Cancer AJCC v8; Stage III Vulvar Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIA Vulvar Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIB Vulvar Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC Vulvar Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVA Vaginal Cancer AJCC v8; Stage IVA Vulvar Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (sexual health counseling) (Experimental): Patients receive sexual health counseling prior to starting and at the completion of radiation.
  Interventions: Other: Counseling; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Counseling — Receive sexual health counseling
  Other Names: Counseling Intervention
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies a sexual health counseling intervention during radiation therapy in improving quality of life for women with gynecologic cancer. Women with gynecologic cancer often suffer long-term complications from treatment that can affect their physical and psychological well-being. An early sexual health counseling intervention prior to and after radiation may improve symptoms management and reduce the physical and psychological effects of treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of a sexual health counseling intervention before and after pelvic radiation for women with gynecologic cancers.

SECONDARY OBJECTIVE:

I. To preliminarily evaluate the efficacy of a sexual health counseling intervention on patient reported outcomes in quality of life, sexual function, and genitourinary symptoms.

OUTLINE:

Patients receive sexual health counseling prior to starting and at the completion of radiation.

After completion of study, patients are followed up at 1 and 6 months after radiation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with endometrial, cervical, vaginal, or vulvar cancer receiving adjuvant external beam radiation or definitive external beam radiation and brachytherapy will be eligible for the study
* Those receiving concurrent chemotherapy will be eligible
* Any prior gynecologic surgery is permitted

Exclusion Criteria:

* Patients with metastatic or recurrent disease and patients receiving brachytherapy alone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Overall completion | Up to 6 months post radiation
  Patients' characteristics and responses to the questionnaires will be summarized using appropriate summary statistics based on their distributions. Parametric tests such as the student's t test and Chi-square test or nonparametric tests such as Mann-Whitney U test and Fisher's exact test will be used to compare patients' characteristics between patients who completed the program and those who did not.
Individual completion of the counseling sessions and questionnaires | Up to 6 months post radiation
  Patients' characteristics and responses to the questionnaires will be summarized using appropriate summary statistics based on their distributions. Parametric tests such as the student's t test and Chi-square test or nonparametric tests such as Mann-Whitney U test and Fisher's exact test will be used to compare patients' characteristics between patients who completed the program and those who did not.

SECONDARY OUTCOMES:
Quality of life (QoL) | Up to 6 months post radiation
  Will be assesses using the European Organization for Research and Treatment of Cancer (EORTC) Core QoL Questionnaire (EORTC QLQ-C30). Data will be displayed graphically using boxplots, histograms and scatterplots to identify interesting features and potential outliers.
Sexual function | Up to 6 months post radiation
  Will be assessed using the EORTC QLQ-CX24. Data will be displayed graphically using boxplots, histograms and scatterplots to identify interesting features and potential outliers.
Genitourinary symptoms using Vaginal Heal Assessment (VHA) | Up to 6 months post radiation
  Will be assessed using the VHA. Data will be displayed graphically using boxplots, histograms and scatterplots to identify interesting features and potential outliers.The Vaginal Health Assessment, the examination tool used in the clinical validation of the VAS, will be utilized to for the gynecologic physical examination for all patients. 15 The assessment evaluates the physical aspect of the vagina including agglutination, adhesions, pH, dryness, rugosity, elasticity, length, thickness, epithelial integrity, vascularity, and irritation. Vaginal diameter will also be assessed during the manual portion of the exam.
  Estimates will be <2.5, 2.5, 3.0, 3.5, 4.0 or >4 cm. 16
Genitourinary symptoms using Vaginal Assessment Scale (VAS) | Up to 6 months post radiation
  Will be assessed using the VAS. Data will be displayed graphically using boxplots, histograms and scatterplots to identify interesting features and potential outliers. Each item is scored from 0 (none) to 3 (severe) and a composite score is calculated by taking the mean of the items.
  A lower score indicates better function. In cancer patients and survivors, the scale were found to have high internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Allison M Quick, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04269837/ICF_000.pdf